CLINICAL TRIAL: NCT07132801
Title: Comparison of Two Qualia NAD⁺ Formulations on Intracellular NAD⁺ Levels: A Randomized, Double-Blind, Placebo-Controlled Three-Arm Trial
Brief Title: Comparison of Two Qualia NAD⁺ Formulations on Intracellular NAD⁺ Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: QLS-014
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: NAD; NAD+ Levels in the Blood
Keywords: NAD Supplementation; NAD

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qualia NAD⁺ version 1 (Active Comparator)
  Interventions: Dietary Supplement: Qualia NAD⁺ version 1
- Qualia NAD⁺ version 2 (Active Comparator)
  Interventions: Dietary Supplement: Qualia NAD⁺ version 2
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Qualia NAD⁺ version 1 — Qualia NAD+ version 1 manufactured by Qualia Life Sciences
  Arms: Qualia NAD⁺ version 1
Dietary Supplement: Qualia NAD⁺ version 2 — Qualia NAD+ version 2 manufactured by Qualia Life Sciences
  Arms: Qualia NAD⁺ version 2
Dietary Supplement: Placebo — Rice Flour
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group study evaluating the effects of two distinct Qualia NAD⁺ formulations on intracellular NAD⁺ levels in healthy adults aged 35-75 years. Approximately 180 participants will be randomized to one of three study arms: Qualia NAD⁺ version 1, Qualia NAD⁺ version 2, or placebo. Each participant will take two capsules of their assigned product once daily in the morning, with or without food, over a 28-day period. The primary outcome is the change in intracellular NAD⁺ levels, assessed via at-home finger-stick blood collection at baseline and study completion. Secondary endpoints include changes in aging-related symptoms (AMFS scores), health-related quality of life (RAND SF-36), and evaluation of safety and tolerability. All assessments, including electronic questionnaires, are completed remotely without in-person visits.

ELIGIBILITY:
Inclusion Criteria:

Provide voluntary, written, informed consent to participate in the study Agree to provide a valid cell phone number and are willing to receive communications through text Can read and write English Willing to not begin taking any new supplements during the study and continue taking any supplements they are currently using regularly Willing to complete questionnaires, records, and diaries associated with the study.

Healthy male and female participants aged 35-75 years Willing to self-administer the intracellular NAD⁺ finger-stick test at home (baseline and Day 28) Willing to avoid supplements, energy drinks/shots, or other products containing niacin, niacinamide, nicotinamide riboside, or NMN for ≥ 2 weeks before baseline and throughout the study

Exclusion Criteria:

Women who are pregnant, breastfeeding, or planning to become pregnant during the trial Known food intolerances/allergy to any ingredients in the product Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, cancer Having had a significant cardiovascular event in the past 6 months Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines On immunosuppressive therapy Individuals who were deemed incompatible with the test protocol Adults lacking capacity to consent

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-13 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Between-group change in intracellular NAD⁺ levels | 28 days
  To assess between-group differences in the change in intracellular NAD⁺ levels from baseline to Week 4 following supplementation with Qualia NAD version 1, Qualia NAD version 2, or placebo.

SECONDARY OUTCOMES:
Aging-Related Symptoms (AMFS scores) | 4 weeks
  To evaluate within-group and between-group differences in the change in Aging Male/Female Symptom (AMFS) total and sub-scale scores.
RAND SF-36 Scale Scores | 4 weeks
  To assess within-group and between-group differences in RAND SF-36 domain scores.
Side effect profile as measured by a custom Safety and Tolerability survey | Week 1, 2, 3, and 4
  To evaluate side effect profiles using a custom Safety and Tolerability survey.
Within-group differences in the change in intracellular NAD⁺ levels | 4 weeks
  To assess within-group differences in the change in intracellular NAD⁺ levels

CONTACTS AND LOCATIONS:
Locations (1):
- Qualia Life Sciences, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No